CLINICAL TRIAL: NCT06018636
Title: Dietary Intake/Patterns, Nutritional Status and Their Association With Growth and Development of Children From Remote, Agropastoral Communities of District Swat, Pakistan
Brief Title: Impact of Diet and Nutrition on Growth and Development in Young Children
Acronym: DIGEST
Status: Recruiting | Type: Observational
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: University of Chester (Other); University of Glasgow (Other); University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Nutrition & Child Development
Record Dates: First submitted 2023-08-06; First posted 2023-08-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Nutrition; Growth; Development; Stunting; Wasting; Obesity; Child Development
Keywords: Nutritional status; Malnutrition; Growth; Cognitive Development; Anthropometry; Agropastoral; remote; rural; Urban
MeSH Terms: conditions — Growth Disorders; Cachexia; Obesity; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Infants and young children residing in agropastoral communities of District Swat, Pakistan
- Group 2: Infant and young children residing in urban areas of district Swat, Pakistan

SUMMARY:
The association between nutrition in early life and its long-term health consequences has long been known. However, there is a scarcity of scientific evidence on how nutritional status affects child growth and development in remote, rural agro-pastoral communities with distinct dietary intake habits, geographical location, socio-economic status, and cultures.

DETAILED DESCRIPTION:
Childhood malnutrition is endemic in Pakistan. However, the agro-pastoral communities of Pakistan are at particularly high risk of childhood malnutrition due to low socioeconomic status, hard-to-reach geographic locations, harsh weather, and frequent natural disasters due to rapid climate change. Furthermore, distinct dietary habits and cultures may also influence child nutritional status and health and development in these communities. The present study aims to assess the dietary intake/patterns, nutritional status, and their association with the growth and development of children from remote, agro-pastoral communities of District Swat, Pakistan.

In this prospective cohort study from Pakistan, infants and young children (n=416) aged ≤ 2 years and residing in agro-pastoral communities of District Swat will be recruited and followed every 12 months for 5 years. An age and gender-matched comparison group of children (n=416) will also be recruited from the more urban areas of District Swat. Data on household socio-economic status, Household Food Insecurity Access Scale (HFIAS), Minimum Dietary Diversity (MDD) of Mothers, Infant and young child feeding practices (IYCF), Complimentary Feeding and Eating practices, and growth and development of the children will be assessed from baseline and every 12 months till the child is 5 years old. Anthropometric assessment including height, weight, mid-upper arm circumference (MUAC), and BMI will also be performed at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Households living in the area from the last two 2 years.
* Households having infants or young children ≤ years.
* Households planning to reside in the same area for the next 1 year.

Exclusion Criteria:

* Children with any co-existent systemic diseases, confirmed from medical records.
* Children on continuous medications for any medical issue.
* Physically or mentally handicapped children

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The target population (infants and young children) residing either in rural, agro-pastoral communities or urban clusters will be recruited from the respective communities. A list of potential participants will be obtained from Extended Program on Immunization (EPI) data of available with local health facilities (Basic Health Unit).
Sampling Method: Probability Sample
Enrollment: 832 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Impact of dietary intake/patterns on Child growth as assessed by body mass index (BMI) | 5 years
  Child growth will be assessed through changes in Body Mass Index (BMI) from baseline and each year till the child is 5 years of age. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared. These data will be categorised further on the basis of the dietary intake patterns of the children as assessed by Infant and Young child feeding practices (IYCF) questionnaire.
Impact of dietary intake/patterns on Child development | 5 years
  Assessment of child development from baseline and each year till the child is 5 years of age. Child development will be assessed by changes in Head circumference and a validated questionnaire (Extended Ages and Stages Questionnaire-3). The EASQ-3 contains 21 questions, targeting child's Communication, Gross motor, Fine motor, Problem solving and Personal-Social skills, each having a total score of 0-60 and cut-off value at 22.77, 41.84, 30.16, 24.62 and 33.71, respectively. Score below the cut-off value indicates possible developmental delays while score slightly above the cut-off value indicates further learning activities and monitoring.
Factors associated with child growth as assessed by changes in BMI | 5 years
  The relationship between child growth and socio-demographic characteristics of the parents, household food insecurity, mother dietary intake (minimum dietary diversity score), and childhood trauma (assessed through Childhood Trauma Scale). CTS is a validated questionnaire containing 16 questions on 04 different aspects trauma i.e., Physical Neglect, Physical Abuse, Emotional Neglect and Emotional Abuse. Total score ranges from 0-80 while 0-20 for each section. Each section has four different cut-off values indicating None, Low, Moderate or Severe neglect/abuse.
Factors associated with child development (based on Head circumference and EASQ-3) | 5 years
  The relationship between child development and socio-demographic characteristics of the parents, household food insecurity, mother dietary intake (minimum dietary diversity score), and childhood trauma (assessed through Childhood Trauma Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shahzad, PhD, Principal Investigator — Khyber Medical University
Locations (1):
- Dr. Muhammad Shahzad, Swat, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramakrishnan U. Prevalence of micronutrient malnutrition worldwide. Nutr Rev. 2002 May;60(5 Pt 2):S46-52. doi: 10.1301/00296640260130731. PMID 12035858
- [Background] Roth DE, Krishna A, Leung M, Shi J, Bassani DG, Barros AJD. Early childhood linear growth faltering in low-income and middle-income countries as a whole-population condition: analysis of 179 Demographic and Health Surveys from 64 countries (1993-2015). Lancet Glob Health. 2017 Dec;5(12):e1249-e1257. doi: 10.1016/S2214-109X(17)30418-7. PMID 29132614
- [Background] Lee A, Cheung CK, Lo K, Keung VM, Mui LW, Tam WWS. Studying Impact of Nutrition on Growth (SING): a prospective cohort for comparing the health outcomes of young children with the dietary quality score. BMJ Open. 2017 Nov 8;7(11):e018380. doi: 10.1136/bmjopen-2017-018380. PMID 29122800